CLINICAL TRIAL: NCT04803734
Title: A Randomized, Single-dose, Open-label, Two-way Crossover Pivotal Study to Assess the Bioequivalence Between Albuterol Sulfate Inhalation Aerosol 108 mcg Per Actuation (MDI, eq. to Albuterol 90mcg/Puff) and Proair HFA (Albuterol Sulfate) Inhalation Aerosol 90 mcg Per Actuation (MDI, eq. to Albuterol 90mcg/Puff) in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Between Albuterol Sulfate Inhalation Aerosol 108 mcg Per Actuation and Proair HFA (Albuterol Sulfate) Inhalation Aerosol 90 mcg Per Actuation in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intech Biopharm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TW20-4502
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Results first posted 2023-09-25 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Albuterol Sulfate inhalation aerosol
  Interventions: Drug: Albuterol Sulfate inhalation aerosol 108mcg per actuation
- Reference Group (Active Comparator): Proair HFA (albuterol sulfate) Inhalation Aerosol
  Interventions: Drug: Proair HFA (albuterol sulfate) Inhalation Aerosol 90 mcg per actuation

INTERVENTIONS:
Drug: Albuterol Sulfate inhalation aerosol 108mcg per actuation — MDI, 2 puffs, single dose, fasting
  Other Names: Albuterol 90mcg/puff
  Arms: Test Group
Drug: Proair HFA (albuterol sulfate) Inhalation Aerosol 90 mcg per actuation — MDI, 2 puffs, single dose, fasting
  Other Names: Albuterol 90mcg/puff
  Arms: Reference Group

SUMMARY:
This study was designed to assess the bioequivalence between the test products (Albuterol Sulfate Inhalation Aerosol 108 mcg Per Actuation) and the reference products (Proair HFA [Albuterol Sulfate] Inhalation Aerosol 90 mcg Per Actuation) in healthy volunteers under fasting conditions. The test product was considered bioequivalent to the reference product if the T/R ln-transformed AUC(0-t), AUC(0-inf), and Cmax were within 80.00-125.00% of those of the reference.

DETAILED DESCRIPTION:
A single-dose, randomized, open-label, two-period, two-sequence, two-treatment, single-centre, crossover bioequivalence study was carried out under fasting conditions in healthy adults, aged 20-60 years. For each period, each subject received a single dose as equivalent to 180 mcg of albuterol of the study drugs according to the pre-determined randomization scheme. Each subject was drawn 22 times over the period of 24 hours. Plasma samples were collected and analyzed for albuterol concentrations by using LC-MS/MS. For each subject, there were 2 dosing periods separated by a 14-day washout period. During the study, standardized meals were provided to all subjects while institutionalized.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers, aged 20-60, inclusive.
2. BMI of 18.0-30.0 kg/m², inclusive. The body weight should be over 50 kg, inclusive. (BMI will be calculated as weight in kilogram [kg]/height in meters² [m²]).
3. Healthy or Non Clinical Significant, according to the medical history, ECG, chest X-ray and physical examination as determined by the Principal Investigator/Sub-Investigator.
4. Systolic blood pressure between 90-139 mmHg, inclusive, and diastolic blood pressure between 50-90 mmHg, inclusive, and pulse rate between 50-100 bpm, inclusive and temperature between 35.0-37.4℃.
5. Screening laboratory values within reference range or NCS as determined by the Principal Investigator/Sub-Investigator.
6. Ability to comprehend and be informed of the nature of the study, as assessed by clinical staff. Capable of giving written informed consent prior to receiving any study medication. Must be able to communicate effectively with clinical staff.
7. Willing to fast for at least 14 hours and to consume standard meals.
8. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
9. Agree not to have a tattoo, body piercing, or other any invasive procedure and blood donation until the end of the study.
10. Never-smokers; or former smokers who have smoked ≥ 100 cigarettes in their lifetime and have not consumed any tobacco or tobacco containing products for at least 12 months prior to screening.
11. Subjects who are non-asthmatic, defined as no clinical history of asthma, allergy or atopy.
12. Able to perform special breathing using nebulizer correctly as per the required standard.
13. Subjects must fulfill at least one of the following:

    * Be surgically sterile for a minimum of 6 months;
    * Post-menopausal for a minimum of 1 year;
    * Agree to avoid pregnancy and use medically acceptable method of contraception from screening day until 30 days after the study ends (last study procedure).

Exclusion Criteria:

1. Known history or presence of any clinically significant hepatic (e.g. active liver disease, hepatic impairment), renal/genitourinary (e.g. renal impairment), gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine (e.g. hypothyroidism), immunological, musculoskeletal (e.g. myopathy, rhabdomyolysis), neurological, psychiatric, dermatological, hematological disease, or any other medical conditions, unless determined as not clinically significant by the Principal Investigator/Sub-Investigator.
2. Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the Principal Investigator/Sub-Investigator.
3. Presence of any significant physical or organ abnormality as determined by the Principal Investigator/Sub-Investigator.
4. A positive test result for any of the following: HIV, Hepatitis B surface antigen, Hepatitis C, drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, opiates, phencyclidine, tetrahydrocannabinol), breath alcohol test. Positive pregnancy test for female subjects.
5. Known history or presence of:

   * Alcohol abuse within one year prior to first drug administration;
   * Drug abuse or dependence;
   * Hypersensitivity or idiosyncratic reaction to albuterol, its excipients, and/or related substances;
   * Allergy to standardized meal provided by site and/or presence of any dietary restrictions;
6. Intolerance to and/or difficulty in blood sampling through venipuncture.
7. Abnormal diet patterns (for any reason) during the 4 weeks preceding the study, including fasting, high protein diets etc.
8. Except for screening procedures, blood donation that results in blood loss of not more than 250 ml in the past 2 months prior to first dosing; blood loss of more than 250 ml within 3 months prior to first dosing.
9. Donation of plasma by plasmapheresis within 7 days prior to first drug administration.
10. Individuals who receives an investigational drug from 2 months prior to first drug administration.
11. Consumption of products containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing and products containing grapefruit and/or pomelo (shown to inhibit cytochrome P450 [CYP] 3A4 activity) within 10 days prior to first drug administration.
12. Use of any medication, including oral multivitamins, herbal and/or dietary supplements within 30 days prior to first drug administration (except topical agents without systemic absorption as determined by the Principal Investigator/Sub-Investigator).
13. Females taking oral or transdermal hormonal contraceptives within 30 days prior to first drug administration.
14. Females having used implanted, injected, intravaginal, or intrauterine hormonal contraceptive within 6 months prior to first drug administration.
15. Individuals having undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by Principal Investigator/Sub-Investigator.
16. Using tobacco products, nicotine products (patches, gum etc.) within 6 months prior to first drug administration.
17. Lactating women.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Kuei Chang, MD, Principal Investigator — Tamshui Mackay Memorial Hospital
Locations (1):
- Tamshui Mackay Memorial Hospital, New Taipei City, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-four subjects were recruited and screened for the eligibility.
Pre-assignment Details: Sixty eligible subjects were randomized in the study.
Groups:
- Albuterol Sulfate Inhalation Aerosol First, Then ProairHFA (Albuterol Sulfate) Inhalation Aerosol: Subjects who were randomized to the sequence of Albuterol Sulfate Inhalation Aerosol first, then ProairHFA (albuterol sulfate) Inhalation Aerosol received an orally inhaled dose of 2 puffs of the test product (Albuterol Sulfate inhalation aerosol 108mcg per actuation) in First Intervention Period 1. After the Washout (14 days) period, subjects received an orally inhaled dose of 2 puffs of the reference product (Proair HFA [albuterol sulfate] Inhalation Aerosol 90 mcg per actuation) in the Second Intervention Period 2.
- Proair HFA (Albuterol Sulfate) Inhalation Aerosol First, Then Albuterol Sulfate Inhalation Aerosol: Subjects who were randomized to the sequence of Proair HFA (albuterol sulfate) Inhalation Aerosol first, then Albuterol Sulfate Inhalation Aerosol received an orally inhaled dose of 2 puffs of the reference product (Proair HFA [albuterol sulfate] Inhalation Aerosol 90 mcg per actuation) in First Intervention Period 1. After the Washout (14 days) period, subjects received an orally inhaled dose of 2 puffs of the test product (Albuterol Sulfate inhalation aerosol 108mcg per actuation) in the Second Intervention Period 2.
Period: Overall Study
Arm/Group | Albuterol Sulfate Inhalation Aerosol First, Then ProairHFA (Albuterol Sulfate) Inhalation Aerosol | Proair HFA (Albuterol Sulfate) Inhalation Aerosol First, Then Albuterol Sulfate Inhalation Aerosol
Started | 30 | 30
Completed | 30 | 28
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Summary of Demographic Data and Baseline Characteristics for All Study Participants.
Arm/Group | All Study Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants] — All the subjects in this study were Taiwanese.
  Participants
    American Indian or Alaska Native | 0
    Asian | 60
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 167.8 (6.8)
Weight [Mean (Standard Deviation); unit: kg] | 65.5 (8.6)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.2 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: The maximal observed plasma concentration of Albuterol Sulfate.
Time Frame: 0 hour (pre-dose), as well as at 2, 5, 10, 15, 20, 30, 45 minutes, and 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
Population: R014, R040, R055, R058 had protocol issues including significantly delayed blood sampling and leakage of drug during dosing. R029 and R058 had pre-dose concentrations > 5% of Cmax. Data of remaining 53 subjects was considered for pharmacokinetic and statistical analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Albuterol Sulfate Inhalation Aerosol: Albuterol Sulfate inhalation aerosol 108 mcg per actuation: MDI, 2 puffs, single dose, fasting
- Proair HFA (Albuterol Sulfate) Inhalation Aerosol: Proair HFA (albuterol sulfate) Inhalation Aerosol 90 mcg per actuation: MDI, 2 puffs, single dose, fasting
Arm/Group | Albuterol Sulfate Inhalation Aerosol | Proair HFA (Albuterol Sulfate) Inhalation Aerosol
Number analyzed (Participants) | 53 | 53
pg/mL | 812.477 (281.148) | 945.456 (359.695)
Statistical Analysis 1: Comparison: Albuterol Sulfate Inhalation Aerosol vs Proair HFA (Albuterol Sulfate) Inhalation Aerosol; Test type: Equivalence — To establish bioequivalence of albuterol under fasting conditions, the 90% confidence interval for the ratio of the geometric means between the products should fall within the FDA defined acceptance range of 80.00%-125.00% interval for ln-transformed Cmax; p = 0.0328, ANOVA; Ratio of geometric least square mean = 0.862, 90% CI 2-sided [0.807 to 0.922]

2. Primary Outcome: AUC(0-t)
Description: Area under the concentration time curve from time zero until the last measurable concentration or last sampling time t, whichever occurs first.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Albuterol Sulfate Inhalation Aerosol | Proair HFA (Albuterol Sulfate) Inhalation Aerosol
Number analyzed (Participants) | 53 | 53
hr*pg/mL | 4806.319 (981.477) | 5090.449 (1053.602)
Statistical Analysis 1: Comparison: Albuterol Sulfate Inhalation Aerosol vs Proair HFA (Albuterol Sulfate) Inhalation Aerosol; Test type: Equivalence — To establish bioequivalence of albuterol under fasting conditions, the 90% confidence interval for the ratio of the geometric means between the products should fall within the FDA defined acceptance range of 80.00%-125.00% interval for ln-transformed AUC(0-t); p < 0.0001, ANOVA; Ratio of geometric least square mean = 0.941, 90% CI 2-sided [0.909 to 0.976]

3. Primary Outcome: AUC(0-inf)
Description: Area under the concentration time curve from time zero to infinity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Albuterol Sulfate Inhalation Aerosol | Proair HFA (Albuterol Sulfate) Inhalation Aerosol
Number analyzed (Participants) | 53 | 53
hr*pg/mL | 5204.806 (1081.862) | 5509.006 (1148.747)
Statistical Analysis 1: Comparison: Albuterol Sulfate Inhalation Aerosol vs Proair HFA (Albuterol Sulfate) Inhalation Aerosol; Test type: Equivalence — To establish bioequivalence of albuterol under fasting conditions, the 90% confidence interval for the ratio of the geometric means between the products should fall within the FDA defined acceptance range of 80.00%-125.00% interval for ln-transformed AUC(0-inf); p < 0.0001, ANOVA; Ratio of geometric least square mean = 0.942, 90% CI 2-sided [0.910 to 0.975]

4. Secondary Outcome: Tmax
Description: Time when the maximal plasma concentration is observed.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Albuterol Sulfate Inhalation Aerosol | Proair HFA (Albuterol Sulfate) Inhalation Aerosol
Number analyzed (Participants) | 53 | 53
hr | 0.929 (1.089) | 0.514 (0.529)

5. Secondary Outcome: T1/2
Description: Terminal elimination half-life, estimated as ln(2)/λ.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Albuterol Sulfate Inhalation Aerosol | Proair HFA (Albuterol Sulfate) Inhalation Aerosol
Number analyzed (Participants) | 53 | 53
hr | 6.928 (1.165) | 6.985 (1.357)

6. Secondary Outcome: Kel(λ)
Description: Terminal elimination rate constant, estimated by linear regression analysis of the terminal portion of the ln-concentration vs. time plot.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Albuterol Sulfate Inhalation Aerosol | Proair HFA (Albuterol Sulfate) Inhalation Aerosol
Number analyzed (Participants) | 53 | 53
1/hr | 0.103 (0.019) | 0.103 (0.021)

7. Secondary Outcome: Mean Residence Time (MRT)
Description: Mean residence time (MRT) is calculated by the area under the first moment curve dividing by area under the concentration time curve.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Albuterol Sulfate Inhalation Aerosol | Proair HFA (Albuterol Sulfate) Inhalation Aerosol
Number analyzed (Participants) | 53 | 53
hr | 8.629 (1.202) | 8.474 (1.455)

ADVERSE EVENTS:
Time Frame: Approximately 16 days for each subject.
Description: The population for safety evaluation was defined as all subjects who took at least one of study drugs. Only AE occurs after first dosing will be analyzed for safety assessment.
Groups:
- Test Group: Albuterol Sulfate inhalation aerosol 108 mcg per actuation: MDI, 2 puffs, single dose, fasting
Arm/Group | Test Group | Reference Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 4/60 | 1/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Group (N=60) | Reference Group (N=58)
Throat infection (Infections and infestations) | 1 | 0
Aspartate aminotransferase (AST) increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Alanine aminotransferase (ALT) increased (Investigations) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT04803734/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT04803734/SAP_001.pdf